CLINICAL TRIAL: NCT00560612
Title: Secondary Prevention With Paroxetine vs. Placebo in Subthreshold Posttraumatic Stress Disorder (PTSD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Durham VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VA IRB# 00993
Record Dates: First submitted 2007-11-19; First posted 2007-11-20 (Estimated); Results first posted 2011-01-25 (Estimated); Last update posted 2019-06-18 (Actual); Status verified 2019-05

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: PTSD; Paroxetine; Subthreshold
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Paroxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Paroxetine (Active Comparator): Paroxetine 10 mg-40 mg or placebo; flexible dosing; 12-week duration.
  Interventions: Drug: Paroxetine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Paroxetine — Paroxetine 10 mg-40 mg or placebo; flexible dosing; 12-week duration.
  Arms: Paroxetine
Drug: Placebo — Placebo: same as paroxetine (active comparator)
  Arms: Placebo

SUMMARY:
The purpose of this study is: 1) To document the effectiveness and tolerability of paroxetine for the treatment of subthreshold posttraumatic stress disorder (PTSD) in veterans in the early post-deployment period; and 2) To determine the potential efficacy of paroxetine in preventing the progression of anxiety symptoms to PTSD and other anxiety disorders, and improving overall veteran function.

DETAILED DESCRIPTION:
See brief summary

ELIGIBILITY:
Inclusion Criteria:

1. Veterans 18-55 years of age
2. Diagnosis of subthreshold PTSD (at least one symptom in PTSD symptom clusters B, C, and D by structured interview; with or without functional impairment exposure to war zone stressors)
3. Written informed consent; and
4. A negative serum pregnancy test for women of childbearing potential.

Exclusion Criteria:

1. Lifetime history of DSM-IV diagnosis of bipolar disorder, schizophrenia or other psychotic disorder, or cognitive disorder due to a general medical condition
2. History of substance dependence within the last 3 months
3. Significant suicide risk or serious suicide attempt within the last year
4. Clinically significant medical condition or laboratory or EKG abnormality
5. Women of childbearing potential who are unwilling to practice an acceptable method of contraception
6. Subjects needing concurrent use of psychiatric medications
7. History of hypersensitivity to paroxetine
8. HADS depression subscale score > 12
9. Failure to respond to an adequate trial of paroxetine (20 mg/day x 8 wks).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2006-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine E Marx, MD, MA, Principal Investigator — Durham VAMC
Locations (1):
- Durham VAMC, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient enrollment at the Durham VA Medical Center occurred from February 2006 until July 2008.
Groups:
- Paroxetine: Week 0: Randomization to paroxetine 10 mg per day for 1 week, Week 1: Paroxetine 10-20 mg/day for 2 weeks (increase to 20 mg/day if tolerating 10 mg/day dose without side effects).
  Week 3: Paroxetine 10-20 mg per day for 2 weeks (increase to 20 mg/day, if tolerating 10 mg/day without side effects and if not already taking 20 mg/day).
  Week 5: Paroxetine 10-30 mg per day for 3 weeks (increase to 30 mg/day if receiving 20 mg/day dose and tolerating without side effects).
  Week 8: Paroxetine 10-40 mg per day for 4 weeks (increase to 40 mg/day if receiving 30 mg/day and tolerating without side effects).
  Week 12: Final study visit (no study medication dispensed).
- Placebo: Week 0: Randomization to placebo for 1 week. Week 1: Placebo for 2 weeks (10-20mg). Week 3: Placebo for 2 weeks (10-20mg). Week 5: Placebo for 3 weeks (10-30mg). Week 8: Placebo for 4 weeks (10-40mg). Week 12: Final study visit (no study medication dispensed).
Period: Overall Study
Arm/Group | Paroxetine | Placebo
Started | 5 | 7
Completed | 5 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paroxetine | Placebo | Total
Number analyzed (Participants) | 5 | 7 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 7 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.3 (4.73) | 35.9 (9.69) | 37.3 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 4 | 6 | 10
Region of Enrollment [Number; unit: participants]
  United States | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinician Administered PTSD Scale (CAPS) Scores
Description: Mean change scores in posttraumatic stress disorder symptoms. Raw scores may range from 0 (no symptoms) to 136 (severe symptoms; score of 136 is based on the first 17 CAPS items administered).
  A reduced CAPS score indicates a reduction in (improvement) PTSD symptoms, while an increase in CAPS score indicates an increase (worsening) in PTSD symptoms. The outcome measure is the change in scores before and after treatment. That is, the baseline and at 12 weeks difference scores.
Time Frame: Change in Scores (12 weeks-Baseline)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paroxetine | Placebo
Number analyzed (Participants) | 5 | 7
Units on a scale | -3.40 (7.37) | -5.00 (6.78)
Statistical Analysis 1: Comparison: Paroxetine vs Placebo; Test type: Superiority; p = 0.7054, t-test, 2 sided

2. Secondary Outcome: Change in Short PTSD Rating Interview Scores
Description: The SPRINT contains 8 questions which are rated on a 0-4 scale (0=not at all; 4=very much). The total score is computed from summing questions #1-8 (range=0-32). The higher the total score, the worse the symptoms. The outcome measure is the change in scores before and after treatment. That is, the baseline and Visit 6 difference scores.
Time Frame: Change in Scores (12 weeks-Baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paroxetine | Placebo
Number analyzed (Participants) | 5 | 7
units on a scale | -3.80 (6.14) | -2.00 (1.15)
Statistical Analysis 1: Comparison: Paroxetine vs Placebo; Test type: Superiority; p = 0.4583, t-test, 2 sided

3. Secondary Outcome: Change in Connor Davidson Resilience Scale Scores
Description: This scale measures resilience. Range of scores (0-100). A score of 0 is suggestive of no resilience, a score of 100 is suggestive of high level of resilience. The outcome measure is the change in scores before and after treatment. That is, the baseline and Visit 6 difference scores.
Time Frame: Change in Scores (12 Weeks-Baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paroxetine | Placebo
Number analyzed (Participants) | 5 | 7
units on a scale | -0.80 (11.67) | -1.29 (9.86)
Statistical Analysis 1: Comparison: Paroxetine vs Placebo; Test type: Superiority; p = 0.7443, t-test, 2 sided

4. Secondary Outcome: Change in Hospital Anxiety and Depression Scale Scores
Description: The total HADS score is presented, which is regarded as a global measure of psychological distress. The total score ranges from 0-42. Each individual question is rated on a 4 point scale (0=absent to 3 =extreme presence). The higher the score, the greater level of psychological distress. The outcome measure is the change in scores before and after treatment. That is, the baseline and Visit 6 difference scores.
Time Frame: Change in Scores (12 Weeks-Baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paroxetine | Placebo
Number analyzed (Participants) | 5 | 7
units on a scale | -3.40 (2.70) | -0.17 (1.80)
Statistical Analysis 1: Comparison: Paroxetine vs Placebo; Test type: Superiority; p = 0.065, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Paroxetine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/7
Other Adverse Events (participants affected / at risk) | 5/5 | 5/7
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paroxetine (N=5) | Placebo (N=7)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Decreased Appetite (General disorders) | 0 (0) | 1 (1)
Decreased Interest in Sex (General disorders) | 1 (1) | 0 (0)
Dermatological (General disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (3)
Disorientation (General disorders) | 0 (0) | 1 (1)
Drowsiness (General disorders) | 0 (0) | 1 (2)
Dry Mouth (General disorders) | 0 (0) | 1 (1)
Excitement/Agitation (General disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 2 (2) | 0 (0)
Hypertension (General disorders) | 0 (0) | 1 (1)
Impaired Sexual Performance (General disorders) | 1 (5) | 0 (0)
Increased Appetite (General disorders) | 0 (0) | 1 (1)
Insomnia (General disorders) | 1 (1) | 1 (1)
Joint Pain/Stiffness (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Nasal Congestion (General disorders) | 1 (1) | 0 (0)
Nausea (General disorders) | 2 (3) | 1 (1)
Restlessness (General disorders) | 2 (2) | 0 (0)
Sweating (General disorders) | 1 (1) | 1 (1)
Syncope/Dizziness (General disorders) | 1 (1) | 1 (1)
Tinnitus (General disorders) | 0 (0) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Vertigo (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes